CLINICAL TRIAL: NCT05624398
Title: Visual Outcomes and Patient Satisfaction in Subjects With Stable Open-angle Glaucoma Undergoing Concurrent Minimally Invasive Glaucoma Surgery and IOL Implantation With an Extended-depth-of-focus IOL
Brief Title: Results of Patients With Glaucoma Undergoing Minimally Invasive Glaucoma Surgery in Conjunction With Cataract Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vold Vision P.L.L.C (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Vivity Protocol 001, Rev A
Record Dates: First submitted 2022-11-06; First posted 2022-11-22 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Glaucoma, Open-Angle; Cataract
Keywords: Glaucoma; Cataract; Microstent; Premium IOL
MeSH Terms: conditions — Glaucoma, Open-Angle; Cataract; Glaucoma

STUDY DESIGN:
Intervention Model Description: Prospective, single-center, single-surgeon, single-arm, descriptive study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Treatment Group (Experimental): Subjects implanted with the Vivity IOL undergoing concurrent implantation of the Hydrus Microstent
  Interventions: Device: Vivity IOL

INTERVENTIONS:
Device: Vivity IOL — Cataract surgery with implantation of the Vivity IOL along with concurrent implantation of the Hydrus Microstent
  Other Names: Hydrus Microstent

SUMMARY:
This study is designed to determine how well patients with glaucoma can see following cataract surgery with a special type of lens called an extended-depth-of-focus (EDOF) lens. This lens is intended to reduced the patients need for glasses following cataract surgery. Patients will also undergo a minimally invasive type of glaucoma surgery using a special type of stent to reduce eye pressure, with the goal of better glaucoma control and the reduction in the need for medications to control eye pressure.

DETAILED DESCRIPTION:
To evaluate the range of vision and patient reported outcomes in subjects implanted with Clareon Vivity IOL undergoing concurrent MIGS with the Hydrus Microstent

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects 45 years of age or older
* A visually significant age-related cataract in both eyes
* Diagnosis of mild OAG

  * VF characteristics consistent with glaucoma with mean deviation not worse than -6.00 dB and without fixation threatening scotoma AND/OR with nerve abnormalities consistent with glaucoma (rim notching, rim thinning, disc hemorrhage, nerve fiber layer loss)
  * Medicated IOP ≤25 mmHg on 1-3 hypotensive medications
* Glaucoma must be judged as stable by investigator based on review of subject medical records

  * Stable VF at least 1 year prior to surgery
  * Stable nerve fiber layer at least 1 year prior to surgery
  * IOP stable on current medication regimen at least 3 months prior to surgery
* Shaffer grade of ≥ III in all angle quadrants
* Potential of best corrected visual acuity at distance in the investigator's judgement of at least 0.1 logMAR (20/25) postoperatively
* Able and willing to comply with follow up visits
* Understands and signs the informed consent
* Both eyes of the subject should undergo surgery within 21 days of each other to ensure adequate timing for final visit window of 90 days ± 21 days post operatively

Exclusion Criteria:

* Previous incisional glaucoma surgery or cilio-ablative surgery
* Prior laser trabeculoplasty within 90 days of surgery
* Pseudoexfoliative, angle closure, uveitic, congenital, traumatic, angle recession, or neovascular glaucoma.
* Moderate glaucoma with VF mean deviation between -6.00 dB and -12.00 dB
* Severe and/or progressive glaucoma defined as

  * VF mean deviation worse than -12.00 dB
  * Consistent worsening of visual field on review of subject medical records
  * Consistent and progressive thinning of nerve fiber layer on review of subject medical records
  * Uncontrolled IOP on maximum glaucoma medications
  * Historically poor IOP control with medical therapy
  * Severe focal notching of the optic nerve rim
  * Expectation for future need of incisional glaucoma surgery
* Ocular pathology or other medical condition which, in the investigator's judgment places the subject at increased risk of complications or significant vision loss during study period
* Ocular pathology that in the investigator's judgment may impact visual acuity postoperatively, i.e., significant ocular surface disease, corneal scarring, blepharitis, epiretinal membrane, macular degeneration, history of significant ocular trauma with sequela, etc.
* Pregnant or breastfeeding women
* Prior refractive surgery e.g., LASIK, RK, PRK, etc.
* Subjects with significant complications during surgical procedure e.g., broken capsule, Hydrus Microstent complication, will be exited from the trial
* Subjects who experience visually significant complications related to the Hydrus Microstent during the study period will be exited from the trial

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2022-12-07 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Mean Photopic Monocular Best Corrected Distance Visual Acuity (DCVA) (4 meters) logMAR | 3 months
  Visual acuity measurement

SECONDARY OUTCOMES:
Mean Photopic Monocular Best Distance Corrected Intermediate Visual Acuity (DCIVA) (66 cm) logMAR | 3 months
  Visual acuity measurement
Mean Photopic Monocular Uncorrected Distance Visual Acuity (UCDVA) (4 meters) logMAR | 3 months
  Visual acuity measurement
Mean Photopic Monocular Uncorrected Intermediate Visual Acuity (UCIVA) (66 cm) logMAR | 3 months
  Visual acuity measurement
Mean Photopic Binocular Best Corrected Distance Visual Acuity (DCVA) (4 meters) logMAR | 3 months
  Visual acuity measurement
Mean Photopic Binocular Best Distance Corrected Intermediate Visual Acuity (DCIVA) (66 cm) logMAR | 3 months
  Visual acuity measurement
Mean Photopic Binocular Uncorrected Distance Visual Acuity (UCDVA) (4 meters) logMAR | 3 months
  Visual acuity measurement
Mean Photopic Binocular Uncorrected Intermediate Visual Acuity (UCIVA) (66 cm) logMAR | 3 months
  Visual acuity measurement
Mean Refractive Spherical Equivalent | 3 months
  Average refractive error or residual spectacle prescription remaining following procedure (diopters)
Mean Absolute Prediction Error | 3 months
  Average prescription remaining compared to preoperative prediction (diopters)
Mean post-op refractive astigmatism and the distribution of post-op refractive astigmatism at ≤0.25D, ≤0.50D, ≤0.75D, and ≤1.00D | 3 months
  Examining the distribution or remaining astigmatism in subjects

OTHER OUTCOMES:
Mean Photopic Monocular Best Distance Corrected Near Visual Acuity (DCNVA) (40 cm) logMAR | 3 months
  Visual acuity measurement
Mean Photopic Monocular Uncorrected Near Visual Acuity (UCNVA) (40 cm) logMAR | 3 months
  Visual acuity measurement
Mean Photopic Binocular Best Distance Corrected Near Visual Acuity (DCNVA) (40 cm) logMAR | 3 months
  Visual acuity measurement
Mean Photopic Binocular Best Corrected Distance Low Contrast Visual Acuity (25%) (4 meters) logMAR | 3 months
  Visual acuity measurement using "faded" letters
Mean Mesopic Binocular Best Corrected Distance Low Contrast Visual Acuity (25%) (4 meters) logMAR | 3 months
  Visual acuity measurement using "faded" letters
Quality of Vision Questionnaire (QoV) | 3 months
  The QoV is a validated questionnaire designed to determine what if any visual disturbances are present following surgery. It consists of a 30-item instrument with 10 possible symptoms rated in each of 3 scales (frequency, severity, and bothersome). Examples of common visual disturbances include glare and halo. This outcome measure can be graded on a linear scale with a higher score being a worse outcome (more visual disturbances). This questionnaire takes approximately 5 minutes to complete.
IOL patient satisfaction (IOLSAT) questionnaire | 3 months
  The IOLSAT is a questionnaire inquiring about the need for eyeglasses, vision without eyeglasses, expectations for needed eyeglasses, and visual satisfaction. It consists of 23 questions, the first 21 based on a Likert scale. Questions 22 asks whether the patient would choose the same lens again and 23 if they would recommend the lens to their family and friends.
Mean preoperative IOP versus postoperative IOP | 3 months
  Comparing intraocular pressure before versus after intervention
Mean preoperative medications versus postoperative medications | 3 months
  Comparing the amount of preoperative glaucoma medications before versus after intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Vold Vision P.L.L.C., Fayetteville, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No
The investigators do not plan to share IPD